CLINICAL TRIAL: NCT03058315
Title: A Prospective Cohort Study With 52 Weeks Follow-up Investigating the Influence of Disease Perception on Functional Outcome Among Patients Referred From General Practice to Secondary Care for Treatment of Low Back Pain.
Brief Title: Disease Perception and Recovery From Low Back Pain
Status: Completed | Type: Observational
Sponsor: Central Jutland Regional Hospital (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Sponsor
Other Study IDs: 6300004
Record Dates: First submitted 2017-02-09; First posted 2017-02-20 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2018-04

CONDITIONS: Low Back Pain
Keywords: Physical activity; Disease perception; Pain beliefs; Disability; Advice
MeSH Terms: conditions — Low Back Pain; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Low back pain patients: Cohort of 800 consecutive low back pain patients, 18 years +, who have been referred from general practice to the secondary sector for further examination and MR scan.

SUMMARY:
The main purpose of the study is to investigate the importance of patients' beliefs regarding staying active despite low back pain, among patients referred from general practice to secondary care treatment in Denmark. It is hypothesised that patients believing that staying active will help them recover will have higher odds of a 30%-improvement in The Roland Morris Disability score after 52 weeks compared to patients disagreeing that staying active will lead to better recovery.

DETAILED DESCRIPTION:
Background: According to international guidelines on low back pain (LBP), advice to stay active should be provided from healthcare professionals to all patients with LBP. However, provision of advice to stay active is reported to be diverse. Some primary care healthcare professionals believe that avoidance of activities and work will help the patient recover. Consequently some patients are not receiving optimal advice to stay active and may think that inactivity will help them and consequently achieve less favourable treatment outcomes. Thus, changing patients' beliefs are considered the key decisive factor to change actual behaviour, and by that improve the functional ability of the patients. This should reduce primary health care use and reduce referrals to the more expensive treatments in secondary care. The effect of patients' beliefs on their functional outcomes has to our knowledge never been studied in a population of patients with LBP being referred from primary care to secondary care treatment.

Materials and Methods:

This is a prospective cohort study. Data is collected from a consecutive series of 800 adult patients (18+), with low back pain as the dominant musculoskeletal complaint, referred from general practices in Central Denmark Region to the Spine Centre at Silkeborg Regional Hospital. Patients will be excluded in case of spinal fractures or malignancy.

All patients seen at the Spine Centre receive a digital letter with a link to an online questionnaire to be completed approximately one week before their appointment at the Spine Centre. The questionnaire contains questions about their back pain history, present pain (Low Back Pain Rating Scale), disability (Rolland Morris Disability Questionnaire), quality of life (EQ-5D), fear-avoidance questions (Örebro Musculoskeletal Pain Questionnaire), STarT Back Screening tool, questions on average level of physical activity, beliefs about physical activity in relation to back pain, advice received from health professionals about staying active, and questions about employment and housing situation. For those accepting participation the same questionnaire is forwarded by email 52 weeks after the initial visit at the Spine Center.

Expected outcome and perspective: This study will bring knowledge about the associations between patient's disease perceptions and beliefs about staying active despite pain and their functional improvement. Furthermore, the study will clarify to what extent patients perceive to have been given advice to stay active by a primary care health professional. Although this study does not explain why some patients do not have guideline concordant beliefs, it will help inform health care professionals in primary care about the possible potential of an increased primary care attention towards the recommendation of staying active when patients have LBP.

ELIGIBILITY:
Inclusion Criteria:

* Low back pain (with or without sciatica) as the dominant musculoskeletal complaint
* 18 years or older

Exclusion Criteria:

* Spinal fractures
* Malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of 800 consecutive low back pain patients referred from primary care to the Spine Centre at Silkeborg Regional Hospital.
Sampling Method: Probability Sample
Enrollment: 828 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Change in Rolland Morris Disability Questionnaire | Change from baseline to 52 weeks
  Validated questionnaire containing 23 questions on self-reported disability due to low back pain

SECONDARY OUTCOMES:
Change in Low Back Pain Rating Scale | Change from baseline to 52 weeks
  Validated questionnaire containing 6 questions on self-reported back and leg pain intensity
Change in EuroQol 5 Dimensions (quality of life) | Change from baseline to 52 weeks
  Validated questionnaire containing 5 questions on self-reported generic quality of life
Change in proportion on sick leave | Change in proportion of patients on sick leave from baseline to 52 weeks
  Self-reported average weekly sick leave during the past 4 weeks
Received consultations in primary sector after referral to secondary care | Measured at 52 week follow-up
  Any consultations with GP, physiotherapist or chiropractors in the year following referral to secondary care due to low back pain (YES/NO)
Change in Major Depression Inventory (depression) | Change from baseline to 52 weeks
  Validated questionnaire containing 10 questions regarding symptoms of depression

CONTACTS AND LOCATIONS:
Overall Officials: Nanna Rolving, PhD, Principal Investigator — Diagnostic Centre, Silkeborg Regional Hospital
Locations (1):
- Diagnostic Centre, Regional Hospital Silkeborg, Silkeborg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bishop A, Foster NE, Thomas E, Hay EM. How does the self-reported clinical management of patients with low back pain relate to the attitudes and beliefs of health care practitioners? A survey of UK general practitioners and physiotherapists. Pain. 2008 Mar;135(1-2):187-95. doi: 10.1016/j.pain.2007.11.010. PMID 18206309
- [Background] Dima A, Lewith GT, Little P, Moss-Morris R, Foster NE, Bishop FL. Identifying patients' beliefs about treatments for chronic low back pain in primary care: a focus group study. Br J Gen Pract. 2013 Jul;63(612):e490-8. doi: 10.3399/bjgp13X669211. PMID 23834886
- [Background] Glasziou P, Haynes B. The paths from research to improved health outcomes. Evid Based Nurs. 2005 Apr;8(2):36-8. doi: 10.1136/ebn.8.2.36. No abstract available. PMID 15830412
- [Derived] Udby CL, Riis A, Thomsen JL, Rolving N. Does the use of telephone reminders to increase survey response rates affect outcome estimates? An ancillary analysis of a prospective cohort study of patients with low back pain. BMC Musculoskelet Disord. 2021 Oct 20;22(1):893. doi: 10.1186/s12891-021-04787-4. PMID 34670521
- [Derived] Riis A, Karran EL, Thomsen JL, Jorgensen A, Holst S, Rolving N. The association between believing staying active is beneficial and achieving a clinically relevant functional improvement after 52 weeks: a prospective cohort study of patients with chronic low back pain in secondary care. BMC Musculoskelet Disord. 2020 Jan 20;21(1):47. doi: 10.1186/s12891-020-3062-6. PMID 31959168